CLINICAL TRIAL: NCT00790894
Title: Phase II Randomized Trial of Ixabepilone Administered Weekly or Every Three Weeks in Patients With HER-2 Negative Metastatic Breast Cancer Previously Treated With Chemotherapy in the Neo-adjuvant or Adjuvant Setting
Brief Title: Trial of Ixabepilone in Patients With HER-2 Negative Metastatic Breast Cancer (HIT)
Acronym: HIT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The low accrual rate of the study (25% of the expected accrual rate)
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: G. Fountzilas/President, Hellenic Cooperative Oncology Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE 11A08
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-05

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: ixabepilone
- 2 (Experimental)
  Interventions: Drug: ixabepilone

INTERVENTIONS:
Drug: ixabepilone — Arm A: ixabepilone will be given at a dose of 40 mg/m2 as a 3-hour intravenous infusion on Day 1 in a 21 days cycle.
  Arms: 1
Drug: ixabepilone — Arm B: ixabepilone will be given at a dose of 20 mg/m2 as a 3-hour intravenous infusion on Days 1, 8 and 15, then 1 week off in a 28-days cycle.
  Arms: 2

SUMMARY:
This is a Phase II Randomized, Open Label, Non-comparative Trial (Parallel Assignment and Efficacy Study) for patients with HER-2 Negative Metastatic Breast Cancer Previously Treated With chemotherapy in the Neo-Adjuvant or Adjuvant Setting.Patients will be randomized to receive Ixabepilone either every three weeks, or weekly for three weeks followed by one week off. Patients will be treated until consent withdrawal, intolerable toxicity or documented disease progression

DETAILED DESCRIPTION:
Patients with measurable metastatic breast cancer that have been treated in the adjuvant or neo-adjuvant setting with chemotherapy will be considered for this study. Subjects must not have received cytotoxic chemotherapy for locally recurrent/metastatic disease. Patients who fulfil the eligibility criteria, and have signed inform consent for the trial will be centrally randomized by electronic means to one of two ixabepilone treatment arms. Stratification factors will include: time to recurrence from adjuvant treatment, calculated from the date of the last dose of adjuvant treatment to the date of relapse (≤ 1 year vs. > 1 year); and previous chemotherapy with taxane regimen in the neo-adjuvant or adjuvant setting (yes vs. no). Randomization will be balanced by site.Treatment Protocol· Arm A [standard once every three weeks schedule]:Ixabepilone [BMS-247550] will be administered on Day 1 (D1) every three weeks as a 3-hour infusion at a dose of 40 mg/m2. · Arm B [weekly schedule]:Ixabepilone [BMS-247550] will be administered weekly for three weeks as a 3-hour infusion at a dose of 20 mg/m2, followed by one week-off.Treatment can be continued until consent withdrawal by the patient, intolerable toxicity or documented disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Female patients aged 18 to 75 years inclusive
* Prior chemotherapy in the adjuvant or neo-adjuvant setting
* Diagnosis of HER-2 negative (HER-2 <2+ by immunohistochemistry and/or FISH negative) metastatic breast adenocarcinoma confirmed by the pathology department of the enrolling institution
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Life expectancy of at least 12 weeks
* Measurable disease by the Response Criteria in Solid Tumors (RECIST) method
* Laboratory values within the specified ranges within 1 week of study enrolment:
* Absolute neutrophil count of ≥ 1.5 x 109/L
* Thrombocyte count of ≥ 100 x 109/L
* Subjects must not have received cytotoxic chemotherapy for locally recurrent/metastatic disease
* Prior hormonal therapy for locally recurrent or metastatic disease allowed
* AST and ALT ≤ 2.5 x ULN
* Bilirubin ≤ 1.5 x ULN
* Recovery from prior palliative radiotherapy for bone metastases

Exclusion Criteria:

* Because of concerns that ixabepilone metabolism may be inhibited by potent cytochrome P450 3A4 inhibitors, patients must not receive the following medications, up to 72 hours prior to initiation of study therapy and until they come off treatment with ixabepilone: amprenavir, delavirdine, voriconazole, erythromycin, cyclosporine, troleandomycin, terfenadine, ketoconazole, nelfinavir, and ritonavir
* Patients with CTC grade 2 or greater neuropathy at baseline
* Patients with any history or evidence of brain an/or leptomenigneal metastasis
* Patients with clinically significant cardiac disease (e.g. unstable angina, congestive heart failure, myocardial infarction) within 6 months from study entry
* Psychiatric disorders or other conditions rendering the subject incapable of complying with the requirements of the protocol
* Any concurrent active malignancy other than non-melanoma skin cancer or in situ carcinoma of the cervix (subjects with a history of previous malignancies but without evidence of disease for 5 years will be allowed to enter the trial)
* Prior severe HSR to agents containing Cremophor EL
* Women of childbearing potential (WOCBP) who are unwilling or unable to use an adequate method of contraception to avoid pregnancy throughout the study and for up to 12 weeks from the last dose of ixabepilone, in such a manner that the risk of pregnancy is minimized WOCBP include: any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea ≥ 12 consecutive months; women on hormone replacement therapy with documented FSH level > 35mIU/mL. Even women who are practising abstinence or whom their partner is sterile (e.g. vasectomy) should be considered of childbearing potential.
* Women who are pregnant or breastfeeding
* Women with a positive pregnancy test on enrolment or prior to study therapy
* No other concomitant chemotherapy, endocrine therapy, immunotherapy, radiation therapy (except for palliative radiotherapy for bone metastases) or investigational treatments are allowed during subject's participation in the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-11; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is the best Overall Response (OR). | At 6, 12 and 24 weeks

SECONDARY OUTCOMES:
Efficacy endpoints: time to response, PFS, TTF, duration of response | Duration of the study
OS Toxicity endpoints: incidence of hematological and non-hematological toxicities | Duration of the study
Translational endpoints | Duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: George Fountzilas, Principal Investigator — Papageorgiou General Hospital
Locations (13):
- Greece (13):
  - Hippokration General Hospital, Oncology Department, Athens
  - University Hospital Attikon, Second Department of Internal Medicine, Oncology Section, Athens
  - Agii Anargiri Cancer Hospital, Third Department of Medical Oncology, Athens
  - Hygeia Hospital, First Deparment of Medical Oncology, Athens
  - Hygeia Hospital, Second Department of Medical Oncology, Athens
  - Alexandra Hospital, Department of Clinical Therapeutics, Athens
  - University General Hospital of Ioannina, Medical Oncology Department, Ioannina
  - University Hospital of Larisa, Department of Medical Oncology, Larissa
  - University Hospital of Patras, Department of Medicine, Division of Oncology, Pátrai
  - Metropolitan Hospital, First Department of Medical Oncology, Piraeus
  - Metropolitan Hospital, Second Dept of Medical Oncology, Piraeus
  - "Theageneio" Cancer Hospital, Third Department of Medical Oncology, Thessaloniki
  - "Papageorgiou" General Hospital, Department of Medical Oncology, Thessaloniki

REFERENCES:
- [Derived] Fountzilas G, Kotoula V, Pectasides D, Kouvatseas G, Timotheadou E, Bobos M, Mavropoulou X, Papadimitriou C, Vrettou E, Raptou G, Koutras A, Razis E, Bafaloukos D, Samantas E, Pentheroudakis G, Skarlos DV. Ixabepilone administered weekly or every three weeks in HER2-negative metastatic breast cancer patients; a randomized non-comparative phase II trial. PLoS One. 2013 Jul 23;8(7):e69256. doi: 10.1371/journal.pone.0069256. Print 2013. PMID 23935969